CLINICAL TRIAL: NCT07023393
Title: Effectiveness of an Intraoperative Spine Measurement Tool and Outcomes Assessment From Its Use in Spinal Fusion Surgery
Brief Title: Proprio Spine Measurement Tool
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Proprio Vision, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00118206
Record Dates: First submitted 2025-06-10; First posted 2025-06-17 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Intervertebral Disc Degeneration; Intervertebral Disc Displacement; Spinal Curvatures; Spinal Osteochondrosis; Spinal Osteophytosis; Spinal Stenosis; Spondylitis; Spondylosis
Keywords: Spine surgery; Proprio; Spine Measurement; Adults; Posterior Spine Surgery; Spine Fusion; Thoracic Spine Surgery; Lumbar Spine Surgery; Sacral Spine Surgery
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral Disc Displacement; Spinal Curvatures; Spinal Osteochondrosis; Spinal Osteophytosis; Spinal Stenosis; Spondylitis; Spondylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Thoracolumbosacral posterior spine surgery using intraoperative measurement system (Experimental): To evaluate the effectiveness of a novel intraoperative spinal measurement tool to assist the surgeon with achieving preoperatively planned alignment-related parameters during surgery. Patients may also be included when the surgeon uses another system or method for placement of the implants (i.e., other navigation system, robot, fluoroscopy, etc.) but also wants to utilize the measurement system. The data will be analyzed as a pool and stratified according to level and # of levels and other demographic and operative data to determine if there are differences.
  Interventions: Device: Intraoperative spinal measurement system

INTERVENTIONS:
Device: Intraoperative spinal measurement system — The design is a prospective study to evaluate the effectiveness of a novel intraoperative spinal measurement tool to assist the surgeon with achieving preoperatively planned alignment-related parameters during surgery.
  Other Names: Paradigm TM System by Proprio

SUMMARY:
This study will prospectively collect data to evaluate the effectiveness of a novel intraoperative spinal measurement system to assist the surgeon with intraoperatively achieving pre-planned alignment-related parameters to the patient's spine. The study will also collect outcomes data to determine if achievement of these spinal alignment-related parameters result in satisfactory outcomes and if it reduces the rate of secondary surgeries.

Objectives

Primary: To evaluate the effectiveness of a novel intraoperative spinal measurement system to assist the surgeon with achieving the surgeon's preplanned alignment-related parameters intraoperatively.

Secondary: To determine if there is a correlation between 1) achievement of preoperative planned alignment-related parameters intraoperatively, and 2) outcomes.

Hypothesis

The application of the intraoperative spinal measurement tool for patients undergoing spinal fusion surgery will improve the surgeon's ability to achieve pre-planned alignment-related parameters intraoperatively and doing so will provide improved outcomes.

DETAILED DESCRIPTION:
Patient reported outcomes data will be collected on two separate forms- the Oswestry Disability Index (ODI) and the SF-36. The ODI has been widely used since its development in 1980 and has been viewed as effective for measuring disability in daily living associated with low back pain4. The SF-36 is the most used patient reported outcomes measure used both generically as well as specifically for low back pain, and it consists of both a mental as well as physical assessment5. Study data will be compared to historical literature data.

The intraoperative spinal measurement system to be used is the Paradigm TM System by Proprio.

Patients will fill out ODI and SF-36 and will have a postoperative standing long x-ray or EOS at regular follow-up intervals (typically 6w, 3m, 6m, 12m, 24m).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older at the time of surgery
* Type of Surgery: Consecutively scheduled patients where the measurement system will be used who will have thoracolumbosacral posterior spine surgery that includes spinal instrumentation and fusion and that consent to the study

Exclusion Criteria:

* Patients treated for traumatic injury (penetrating injuries, etc.)
* Incarcerated persons
* Pregnant females
* Any patient current in another trial for a new implant or technique
* Non-Spine Related Surgeries: Patients who had surgeries for reasons other than spine-related conditions (even if they incidentally involved the spine)
* Patients having additional surgery occurring concurrently with spine surgery
* Patients ineligible for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2027-02-05 (Estimated); Study Completion 2029-02-05 (Estimated)

PRIMARY OUTCOMES:
Number of times the adjustment tool failed to represent the POF within a margin of 3 degrees | Pre-operative planned state (enrollment), Postoperative final state (12 months)
  Effectiveness of the intraoperative spinal measurement tool will be assessed

SECONDARY OUTCOMES:
Patient Reported Outcomes as measured by the Oswestry Disability Index (ODI) | Enrollment to 24 months post-operatively
  The Oswestry Disability Index (ODI) measures disability in daily living associated with low back pain. The total score is calculated as a percentage, with 0% indicating no disability and 100% indicating the highest level of disability.
Patient Reported Outcomes as measured by the 36-Item Short Form Survey (SF-36) | Enrollment to 24 months post-operatively
  The SF-36 measures health-related quality of life across eight domains, each scored 0-100 (higher = better health). Two summary scores-Physical Component Summary (PCS) and Mental Component Summary (MCS)-are derived.
Number of secondary surgeries | Enrollment to 24 months post-operatively
  Number of secondary surgeries will be collected through the electronic health record and from the patient to capture any surgery performed outside Duke.

CONTACTS AND LOCATIONS:
Overall Officials: Brett Rocos, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finkelstein JA, Schwartz CE. Patient-reported outcomes in spine surgery: past, current, and future directions. J Neurosurg Spine. 2019 Aug 1;31(2):155-164. doi: 10.3171/2019.1.SPINE18770. Epub 2019 Aug 1. PMID 31370009
- [Background] Beighley A, Zhang A, Huang B, Carr C, Mathkour M, Werner C, Scullen T, Kilgore MD, Maulucci CM, Dallapiazza RF, Kalyvas J. Patient-reported outcome measures in spine surgery: A systematic review. J Craniovertebr Junction Spine. 2022 Oct-Dec;13(4):378-389. doi: 10.4103/jcvjs.jcvjs_101_22. Epub 2022 Dec 7. PMID 36777909
- [Background] Lau KKL, Samartzis D, To NSC, Harada GK, An HS, Wong AYL. Demographic, Surgical, and Radiographic Risk Factors for Symptomatic Adjacent Segment Disease After Lumbar Fusion: A Systematic Review and Meta-Analysis. J Bone Joint Surg Am. 2021 Aug 4;103(15):1438-1450. doi: 10.2106/JBJS.20.00408. PMID 34166276
- [Background] Radcliff KE, Kepler CK, Jakoi A, Sidhu GS, Rihn J, Vaccaro AR, Albert TJ, Hilibrand AS. Adjacent segment disease in the lumbar spine following different treatment interventions. Spine J. 2013 Oct;13(10):1339-49. doi: 10.1016/j.spinee.2013.03.020. Epub 2013 Jun 15. PMID 23773433
- [Background] Ikard RW. Methods and complications of anterior exposure of the thoracic and lumbar spine. Arch Surg. 2006 Oct;141(10):1025-34. doi: 10.1001/archsurg.141.10.1025. PMID 17043282